CLINICAL TRIAL: NCT03952104
Title: Effects of Different Strength Training Programs on Quality of Life in Elderly
Brief Title: Strength Training and Quality of Life in Elderly
Acronym: ST-QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-19
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Quality of Life
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental-Low Intensity Strength Training (Experimental): Strength training (low intensity)
  Interventions: Other: Strength training
- Experimental-Moderate Intensity Strength Training (Experimental): Strength training (moderate intensity)
  Interventions: Other: Strength training
- Experimental-High Intensity Strength Training (Experimental): Strength training (high intensity)
  Interventions: Other: Strength training
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Strength training — Strength training
  Arms: Experimental-High Intensity Strength Training; Experimental-Low Intensity Strength Training; Experimental-Moderate Intensity Strength Training

SUMMARY:
Aim: To evaluate the impact of three different strength training programs on psychological wellbeing of elderly.

DETAILED DESCRIPTION:
Background: Physical activity in the elderly has benefits which improve psychological wellbeing. However, the majority of older adults perform less physical activity with advancing age.

Aim: To evaluate the impact of three different 32-week strength training programs (low, moderate and high intensity) on psychological wellbeing of elderly.

Design: Randomized Controlled Trial.

ELIGIBILITY:
Inclusion Criteria:

* age ≥60 years;
* having the ability to speak and write in Spanish;
* having the ability to complete the questionnaires independently.

Exclusion Criteria:

-the presence of any medical problem or pathology that could hinder physical activity practice

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Quality of life, assessed through the Short Form 36 health survey questionnaire. | 32 weeks
  This questionnaire measures quality of live. It provides information on 8 scales, scoring from 0 (worst health) to 100 (best health), and on the physical component scale (PCS) and the mental component scale (MCS), normalized scores representing overall physical and mental functioning.

SECONDARY OUTCOMES:
Emotional wellbeing, assessed through the STAI (State-Trait Anxiety Inventory) questionnaire. | 32 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress. STAI has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Motivation towards physical activity, assessed through the Behavioural Regulation in Exercise Questionnaire (BREQ-2) | 32 weeks
  This questionnaire consists of 19 items measuring stages on the continuum of self-determination. It measures external regulation (4 items), introjected regulation (3 items), identified regulation (4 items), intrinsic regulation (4 items), and it adds amotivation (4 items) on a scale from 1 (Not at all true for me) to 5 (Absolutely true for me). Each of the subscales has a maximum score, with a maximum of 20 for external regulation, identified regulation, intrinsic regulation and amotivation, and 15 for introjected regulation.

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, PhD, Study Director — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain